CLINICAL TRIAL: NCT02986022
Title: A Psychological Intervention to Enhance Resilience in Mainland New Immigrants to Hong Kong
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City University of Hong Kong (Other)
Collaborators: International Social Service Hong Kong Branch (Unknown)
Responsible Party: Principal Investigator, Nancy Xiaonan Yu, Assistant Professor, City University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCPF2016
Record Dates: First submitted 2016-11-29; First posted 2016-12-07 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Resilience
Keywords: Self-efficacy; optimism; altruism; goal setting
MeSH Terms: conditions — Altruism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resilience (Experimental): Participants will receive four sessions covering Resilience intervention content
  Interventions: Behavioral: Resilience
- Resilience+Information (Active Comparator): Participants will receive four sessions covering Resilience intervention and Information intervention contents.
  Interventions: Behavioral: Resilience; Behavioral: Information

INTERVENTIONS:
Behavioral: Resilience — Self-efficacy, optimism, altruism, goal setting
Behavioral: Information — Information and resources about education, medical care, housing, employment, and community facilities available in Hong Kong and Mainland China
  Arms: Resilience+Information

SUMMARY:
Background:

Resilience is important for successful adaptation. The investigators' resilience intervention was effective in enhancing resilience, emotional functioning, and adaptation in Mainland immigrants. In the present proposal, the investigators will work with the International Social Service to scale up application of this intervention in immigrants, and develop the training infrastructure to ensure that the evidence-based intervention can be sustained despite turnover of interventionists.

Objectives:

1. We will conduct a randomized controlled trial to compare the resilience intervention with the resilience + information intervention (a compound module) among 200 new immigrants,
2. The resilience intervention will enhance participants' resilience by 5%, and decrease their depressive symptoms by 20% and adaptation difficulties by 10% after the completion of the intervention,
3. The resilience + information intervention will have higher increases in resilience and more decreases in depressive symptoms and adaptation difficulties compared to the resilience intervention, and
4. To establish a sustaining mechanism which ensures that these two interventions can continue to be used in routine services.

Project design:

Well-trained social workers will deliver the intervention. Participants will complete programme evaluation. A train-the-trainer workshop and training materials will be prepared to transfer knowledge to social workers who are future trainers.

DETAILED DESCRIPTION:
The intervention programme has been developed, manualized, and rigorously tested in our previous study (1). This programme is largely a replica of our original programme. Two social workers will deliver the resilience intervention. One of the two interventionists who delivered the intervention in our empirical study is still available. One more social worker will be selected from recently trained interventionists to deliver this intervention.

This resilience intervention (see Supplement 2) consists of 4 sessions, each lasting for 2 hours, finished within two weeks. This intervention is built on the international and local evidence about positive characteristics that promote successful immigration and effective strategies that enhance psychological well-being.

We will promote this intervention programme in new immigrants, and recruit participants by open recruitment, contacting current service users of the community agency, referral and cold call. Orientation gatherings will be organized to screen for eligible immigrants.

The resilience + information intervention consists of 4 sessions, each lasting for 2.5 hours, finished within two weeks. In each session, the resilience section will last for 2 hours (identical to the resilience intervention), and the information intervention will be half an hour. Similar to our previous information intervention, this information section will cover transportation, housing, medical service, education, and employment, the important information helpful for the immigrants' adaptation.

Participants will receive four sessions, either the resilience intervention or the resilience + information intervention. Unlike most programmes that have not been developed in the community, we have identified some key strategies to reduce attrition during the intervention. Before each session, social workers will call participants to remind them of the coming session. During the intervention, we will provide child care upon participants' request. For those who are unable to attend a specific sessions, social workers will conduct a make-up on the content, and provide general encouragement that attendance of further sessions will bring important gains. During the follow-up period, social workers will send reminder postcards to participants. At the end of the intervention, participants will obtain a certificate in recognition of their participation in this programme. Evaluation will be conducted before the first session (pre-intervention) and immediately after the intervention (post-intervention).

ELIGIBILITY:
Inclusion Criteria:

* Immigrants who arrived in Hong Kong from Mainland China less than 3 years ago
* have least a primary school education

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2016-12-07 (Actual); Primary Completion 2018-02-08 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Resilience as assessed by Connor-Davidson Resilience Scale | 1 month

SECONDARY OUTCOMES:
Depressive symptoms as assessed by Patient-Health Questionnaire-9 | 1 month
Adaptation difficulties as assessed by Sociocultural Adaptation Scale | 1 month
Knowledge measured using the items developed in our previous study | 1 month
  Knowledge on services and resources regarding transportation, housing, medical service, education, and employment

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Xiaonan Yu, Principal Investigator — City University of Hong Kong
Locations (1):
- City University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No